CLINICAL TRIAL: NCT06043908
Title: The Effect of Topical 0.05% Cyclosporine Eye Drops on Post-refractive Surgery Dry Eye
Brief Title: The Effect of 0.05% CsA Eye Drops on Post-refractive Surgery Dry Eye
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RS01
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Dry Eye
Keywords: dry eye, refractive surgery, 0.05% cyclosporine
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.05% cyclosporine eyedrops combined with artificial tear eyedrops (Experimental): 0.05% cyclosporine eyedrops combined with artificial tear eyedrops
  Interventions: Drug: artificial tear eyedrops; Drug: 0.05% cyclosporine eyedrops
- artificial tear eyedrops (Active Comparator): artificial tear eyedrops
  Interventions: Drug: artificial tear eyedrops

INTERVENTIONS:
Drug: artificial tear eyedrops — The intervention group and control group were treated with artificial tear eyedrops four times a day.
Drug: 0.05% cyclosporine eyedrops — The intervention group was treated twice a day.
  Arms: 0.05% cyclosporine eyedrops combined with artificial tear eyedrops

SUMMARY:
The purpose of this study is to observe the effect of 0.05% cyclosporine eyedrops combined with artificial tears in patients with dry eyes after corneal refractive surgery and to observe the changes in ocular surface characteristics and tear inflammatory cytokines before and after treatment.

DETAILED DESCRIPTION:
The purpose of this study is to observe the effect of 0.05% cyclosporine eyedrops combined with artificial tears in patients with dry eyes after corneal refractive surgery and to observe the changes in ocular surface characteristics and tear inflammatory cytokines before and after treatment. At the same time, this study further observed whether 0.05% cyclosporine eyedrops combined with artificial tear eyedrops were more beneficial to ocular surface repair and tear film homeostasis compared with traditional artificial tears alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients who suffering from dry eye after refractive surgery with age between 18 and 45 years old.
* Any gender.
* Provision of written informed consent.

Exclusion Criteria:

* active ocular infection, ocular inflammation, active ocular allergy, severe blepharitis or obvious inflammation of the eyelid margin.
* Pregnant and lactating women, or those planning a pregnancy over the course of the study.
* Uncontrolled systemic disease.
* Suffer from diseases that may affect corneal nerves, such as keratoconus, trigeminal neuralgia, allergic conjunctivitis, etc.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
ocular surface disease index (OSDI) | from baseline to 3 months after treatment
  OSDI is one of the most frequently used questionnaires for evaluation of dry eye disease (DED). This includes 12 questions which measure the frequency of symptoms over the recent week, and the scores range from 0 to 100.
Tear break-up time (TBUT)(s) | from baseline to 3 months after treatment
  BUT is the time from normal blinking to the first appearance of a break in the tear film.
Corneal fluorescein staining (CFS) | from baseline to 3 months after treatment
  The degree of fluorescein staining of the cornea was evaluated using the National Eye Institute (NEI) scale of five corneal regions (central, superior, temporal, nasal, and inferior). The scores range from 0 to 15.
Schirmer I test (SIt) (mm/5 minutes) | from baseline to 3 months after treatment
  The Schirmer I test is performed using sterile strips without anesthesia. The strips are placed in the lateral part of the inferior fornix of the eye for 5min and the extent of tear flow down was measured in millimeters.
Lissamine green staining | from baseline to 3 months after treatment
  To grade the temporal zone, the subject looks nasally; to grade the nasal zone the subject looks temporally. The upper and lower conjunctiva can also be graded.

SECONDARY OUTCOMES:
the concentration of Interleukin-1β (IL-1β) (pg/ml) | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-1β levels will be quantified by Luminex immunoassay.
the concentration of Interleukin-6 (IL-6) (pg/ml) | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-6 levels will be quantified by Luminex immunoassay.
the concentration of Interleukin-10 (IL-10) (pg/ml) | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-10 levels will be quantified by Luminex immunoassay.
the concentration of Interleukin-23 (IL-23) (pg/ml) | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-23 levels will be quantified by Luminex immunoassay.
the concentration of Interleukin-17A (IL-17A) (pg/ml) | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-17A levels will be quantified by Luminex immunoassay.
the concentration of tumor necrosis factor-α (TNF-α)(pg/ml) | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. TNF-α levels will be quantified by Luminex immunoassay.
the concentration of interferon-γ (IFN-γ)(pg/ml) | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IFN-γ levels will be quantified by Luminex immunoassay
the concentration of granulocyte-macrophage colony-stimulating factor (GM-CSF)(pg/ml) | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. GM-CSF levels will be quantified by Luminex immunoassay.
the concentration of substance P (SP)(pg/ml) | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this neuropeptide. SP levels will be quantified by Luminex immunoassay.
the concentration of alpha-melanocyte-stimulating hormone (α-MSH) (pg/ml) | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this neuropeptide. α-MSH levels will be quantified by Luminex immunoassay.
the concentration of β-endorphin (pg/ml) | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this neuropeptide. β-endorphin levels will be quantified by Luminex immunoassay
the concentration of neurotensin (pg/ml | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this neuropeptide. β-endorphin levels will be quantified by Luminex immunoassay.
the concentration of oxytocin(pg/ml) | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this neuropeptide. oxytocin levels will be quantified by Luminex immunoassay.
corneal sensitivity (range, 60-0 mm) | from baseline to 3 months after treatment
  Corneal sensitivity will be measured in the right eye only using the Cochet-Bonnet aesthesiometer and the ascending method of limits to determine the threshold of stimulus detection.
sub-basal corneal nerve density (mm/mm2) | from baseline to 3 months after treatment
  Sub-basal corneal nerve plexus image will be acquired using a laser scanning confocal microscope.
numerical rating scale (NRS) | from baseline to 3 months after treatment
  The NRS was used to evaluate ocular pain and consists of a numbered line from 0 to 10 scores that measures pain intensity: 0-1: no pain; 2-4: mild pain; 5-7: moderate pain; and 8-10: severe pain.
NPSI-Eye (range 0-100 score) | from baseline to 3 months after treatment
  Neuropathic Pain Symptom Inventory modified for the Eye (NPSI-Eye) (range 0-100 over a 24-hour recall period)

CONTACTS AND LOCATIONS:
Overall Officials: Hong Qi, Principal Investigator — Peking University Third Hospital
Locations (1):
- Hong Qi, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhao L, Chen J, Duan H, Yang T, Ma B, Zhou Y, Bian L, Cai X, Qi H. Efficacy of topical 0.05% cyclosporine A and 0.1% sodium hyaluronate in post-refractive surgery chronic dry eye patients with ocular pain. BMC Ophthalmol. 2024 Jan 22;24(1):28. doi: 10.1186/s12886-024-03294-z. PMID 38247010